CLINICAL TRIAL: NCT04701580
Title: Longitudinal Measurement of Synaptic Density to Monitor Progression of Huntington's Disease.
Brief Title: Synaptic Density and Progression of Huntington's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s61478
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; PET; 11C-UCB-J; 18F-FDG; SV2A
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: Longitudinal study design (2 years follow up) where results of SV2A PET/CT, FDG PET/MR and clinical rating scales are compared between HD patients and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD patients (Experimental): At baseline and 2-year follow-up
  Interventions: Diagnostic Test: 11C-UCB-J PET-CT; Diagnostic Test: 18F-FDG PET-MR
- Healthy controls (Active Comparator): At baseline and 2-year follow-up
  Interventions: Diagnostic Test: 11C-UCB-J PET-CT; Diagnostic Test: 18F-FDG PET-MR

INTERVENTIONS:
Diagnostic Test: 11C-UCB-J PET-CT — Positron Emission Tomography (PET) of synaptic vesicle protein 2A (SV2A) using the radioligand 11C-UCB-J.
Diagnostic Test: 18F-FDG PET-MR — Positron Emission Tomography (PET) of glucose metabolism using the radioligand 18F-FDG, and brain MRI performed simultaneously.

SUMMARY:
AIM: To assess synaptic density and to investigate the potential relationship of regional synaptic loss with motor and non-motor symptoms and with disease progression in the human brain in vivo in patients with HD.

DESIGN: The investigators will include 20 HD mutations carriers and 15 healthy controls. All subjects will undergo a clinical examination, with comprehensive assessment of motor and non-motor symptoms, and imaging evaluation consisting of 11C-UCB-J PET-CT and 18F-FDG PET-MR at baseline and after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years.
* Capacity to understand the informed consent form.
* For HD group: CAG repeat expansion in HTT ≥ 40.
* Premanifest HD mutation carriers:

  * No clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score < 4.
* Early manifest HD patients:

  * Clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score = 4.
  * UHDRS-TFC score 7 or higher (Shoulson-Fahn stage 1 and 2).

Exclusion Criteria:

* neuropsychiatric diseases other than HD
* major internal medical diseases
* white matter lesion load on FLAIR Fazekas score 2 or higher or other relevant MRI abnormalities
* history of alcohol abuse or current alcohol abuse (chronic use of more than 15 units per week) or drug abuse
* contraindications for MR
* pregnancy
* previous participation in other research studies involving ionizing radiation with >1 mSv in the previous 12 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Baseline differences in synaptic density. | Data analysis wel be done when all subjects have undergone the baseline evaluation.
  Baseline differences (%) in (regional) synaptic density between patients and controls.
Baseline correlations between clinical scores and regional synaptic density. | Data analysis wel be done when all subjects have undergone the baseline evaluation.
  Correlations between clinical scores and regional synaptic density in the patient group at baseline.
Differences in the rate of decline of synaptic density. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Differences (%) in the rate of decline of synaptic density between patients and controls.
Correlations between progression of the clinical scores and decline of synaptic density. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between progression of the clinical scores and decline of synaptic density in the patient group, after longitudinal follow up of 2 years.

SECONDARY OUTCOMES:
Baseline differences in cerebral glucose metabolism. | Data analysis wel be done when all subjects have undergone the baseline evaluation.
  Baseline differences (%) in (regional) glucose metabolism between patients and controls.
Baseline correlations between clinical scores and cerebral glucose metabolism. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between clinical scores and cerebral glucose metabolism in the patient group at baseline.
Differences in the rate of decline of cerebral glucose metabolism. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Differences (%) in the rate of decline in cerebral glucose metabolism between patients and controls.
Correlations between progression of the clinical scores and decline of cerebral glucose metabolism in the patient group, after longitudinal follow up of 2 years. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between progression of the clinical scores and decline of cerebral glucose metabolism in the patient group, after longitudinal follow up of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Vandenberghe, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Needs to be decided.